CLINICAL TRIAL: NCT00399009
Title: Comparative Study of Circular Stapling Instruments Concerning the Risk of Anastomotic Dehiscence After Anterior Resection for Rectal Cancer.
Brief Title: Comparative Study of Circular Stapling Instruments
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: One of the instruments in the study was withdrawn from the market before the calculated number of persons were included.
Sponsor: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ups03-130
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2008-06-09 (Estimated); Status verified 2008-06

CONDITIONS: Anastomotic Leak; Rectal Cancer
Keywords: Circular stapling devices; anastomotic leak; anastomotic dehiscence; rectal cancer
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms

INTERVENTIONS:
Device: AutoSuture Premium Plus CEEA/Ethicon Proximate ILS

SUMMARY:
After removing the rectum at surgery, bowel continuity can sometimes be restored by an anastomosis between the anus and the bowel. This anastomosis is most commonly created by the use of surgical circular stapling instruments. In a retrospective pilot study the risk of developing an acute leak in the anastomosis was increased with one of the most commonly used instruments in Sweden as compared to the other brand in use. In the current study the patient is randomized to either one of the instruments after a resection of the rectum for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Anterior resection for Rectal Cancer
* Informed consent

Exclusion Criteria:

* Can not give informed consent
* Patient can not be followed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Clinical anastomotic leak

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Folkesson, M.D Ph.D., Principal Investigator — Uppsala University; Lars Påhlman, Professor M.D. Ph.D., Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Folkesson J, Brown SS, Gunnarsson U, Pahlman L. Randomised multicentre trial of circular stapling devices. Int J Colorectal Dis. 2012 Feb;27(2):227-32. doi: 10.1007/s00384-011-1307-4. Epub 2011 Sep 10. PMID 21909698